CLINICAL TRIAL: NCT06714435
Title: Effect of Intermittent Hypoxia on Ventilatory Endurance in Healthy Volunteers
Acronym: ENDUR-HYPOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ENDUR-HYPOX
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Intermittent Hypoxia; Respiratory Endurance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe 1 (Experimental): Control visit in normoxia at V1 and then test visit in intermittent hypoxia at V2
  Interventions: Other: Intermittent hypoxia; Other: Normoxia
- Groupe 2 (Experimental): Test visit in intermittent hypoxia at V1 and then control visit in normoxia at V2
  Interventions: Other: Intermittent hypoxia; Other: Normoxia

INTERVENTIONS:
Other: Intermittent hypoxia — Intermittent hypoxia during 6 hours in daytime
Other: Normoxia — Normoxia during 6 hours in daytime

SUMMARY:
Sleep apnoea syndrome is a common disorder responsible for poor sleep quality and repeated oxygen depletion in the blood. Patients suffering from this disease experience a reduction in their endurance, i.e. their ability to make prolonged efforts. This loss of muscular endurance affects breathing in particular. It is known that poor sleep reduces endurance, but it is not knwon whether the repeated lack of oxygen for several hours at night also has this effect. This information could help improve the management of certain acute respiratory illnesses (asthma attacks, respiratory infections, etc.).

This project therefore seeks to establish a link between repeated oxygen deprivation and a reduction in the human brain's ability to train respiratory muscles. To this end, the healthy volunteers in this study will perform the same breathing exercise (breathing for as long as possible through a mask that makes inspiration difficult) twice: once after 6 hours' exposure to repeated oxygen deprivation, and once under conditions of normal oxygenation. The order of these exercises will be randomized. These exercises will take place in a special room, a hypoxia chamber, where it is possible to deplete the air breathed in oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Non-excessive coffee drinker (< 3 espressos / day)
* Non-smoker or weaned for 3 months and total consumption < 10 packs/year
* With a BMI within ]18 - 25[ kg/m².
* Benefiting from a Social Security plan or benefiting from one through a third party
* Giving free, informed and signed consent, after receiving clear and fair information about the study.

Non-inclusion Criteria:

* History of respiratory or ENT disease (asthma, chronic bronchitis, COPD, respiratory allergy, swallowing disorders, oropharyngeal malformation, obstructive or central sleep apnea-hypopnea syndrome, alveolar hypoventilation syndrome)
* Respiratory, cardiovascular, muscular, neurological or diabetic pathology or disorders
* Raynaud's disease/syndrome
* History of epilepsy or history of malaise suggestive of epilepsy
* Psychiatric history requiring hospitalization
* Liver failure
* Renal insufficiency
* History of acute mountain sickness (presence during or after a stay at altitude of symptoms of vertigo, headache, nausea/vomiting and incapacitating fatigue: Lake Louise score > 0)
* History of migraines
* Taking medications that interfere with respiratory function or cardiovascular function, or psychotropic drugs ( anxiolytic, sedative, antidepressant, neuroleptic, muscle relaxant, etc.).
* Alcohol or drug dependence
* Anemia, sickle-cell anemia
* SpO2 < 97% at rest in room air
* Currently participating in another clinical study
* Protected persons within the meaning of article L1121-5 to 8 (persons benefiting from enhanced protection, i.e. minors, persons deprived of their liberty by a judicial or administrative decision, pregnant or breast-feeding women, persons staying in a health or social establishment, adults under legal protection, and patients in emergency situations). - Women with childbearing capacity who do not have effective contraception (hormonal/mechanical: oral, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy).
* Incidental finding of acute mountain sickness (Lake Louise score >0)
* Pregnant woman (incidental finding)
* Persistence of average sleep time < 6h
* Non-reversible deterioration in volunteer's state of health within study period
* Electroencephalogram signal unusable

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
To compare the inspiratory endurance of healthy volunteers after 6h of continuous breathing in room air and after 6h of continuous exposure to intermittent hypoxia in a hypoxic chamber. | through study completion, an average of 2 years

SECONDARY OUTCOMES:
After 6 h of continuous breathing in room air and after 6 h of continuous exposure to intermittent hypoxia in a hypoxic chamber, compare Maximum Inspiratory Pressure (PImax) before and after the inspiratory endurance test. | through study completion, an average of 2 years
Compare inspiratory cortical control measured by EEG over the first 15 and last 15 minutes of the inspiratory endurance test after 6 h of continuous breathing in room air and after 6 h of continuous exposure to intermittent hypoxia in a hypoxic chamber. | through study completion, an average of 2 years
  The inspiratory cortical control is recorded by electroencephalography to measure the amplitude of inspiratory premotor potentials in µV
Compare respiratory discomfort with a visual analog scale at the start of the endurance test after 6 h of continuous breathing in room air and after 6 h of continuous exposure to intermittent hypoxia in a hypoxic chamber. | through study completion, an average of 2 years
  The visual analogue scale ranges from 0 to 10, with 10 being the most severe discomfort
Compare the time to onset of respiratory discomfort in the inspiratory endurance test with a visual analog scale after 6 h of continuous breathing in room air and after 6 h of continuous exposure to intermittent hypoxia in a hypoxic chamber. | through study completion, an average of 2 years
  The visual analogue scale ranges from 0 to 10, with 10 being the most severe discomfort. The time to onset of respiratory discomfort is defined by the time it takes to reach 80% of the maximum discomfort declared by the volunteer.
Compare sensory perception of inspiratory effort after 6 h of continuous breathing in room air and after 6 h of continuous exposure to intermittent hypoxia in a hypoxic chamber. | through study completion, an average of 2 years
Compare the quantity and phenotype of circulating microvesicles in ambient air or in intermittent hypoxia. | through study completion, an average of 2 years
Compare systolic pulmonary artery pressure in room air or intermittent hypoxia using trans-thoracic echography. | through study completion, an average of 2 years
  The systolic pulmonary artery pressure is measured by the following measurements :
  * The maximum regurgitation velocity of tricuspid insufficiency will be measured by continuous Doppler in order to estimate the pressure gradient between the right atrium and the pulmonary artery using Bernoulli's equation.
  * The pressure in the right atrium will be estimated by measuring the diameter of the inferior vena cava and its compliance.
Compare echographic signs of right ventricular function in room air or intermittent hypoxia using trans-thoracic echography. | through study completion, an average of 2 years
  Right ventricular function is estimated by measuring the tricuspid annular plane systolic excursion (TAPSE) and the S wave.

OTHER OUTCOMES:
To compare the somnolence of healthy volunteers after 6h of continuous breathing in room air and after 6h of continuous exposure to intermittent hypoxia in a hypoxic chamber. | through study completion, an average of 2 years
  Number of micro-sleep episodes of at least 3 seconds (stages N1, N2, N3, REM) identified in EEG tracings recorded under both conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Céline ABONNEAU, Study Chair — CHU Poitiers
Locations (1):
- CHU Poitiers, Poitiers, France, France